CLINICAL TRIAL: NCT03018093
Title: A Phase I Study Evaluating Safety and Efficacy of CBM.CD19-targeted Chimeric Antigen Receptor T Cells (C-CAR011) Treatment in Adult Subjects With Relapsed/Refractory CD19+ B Cells Acute Lymphoblastic Leukemia(CALL-1)
Brief Title: A Phase I Study Evaluating Safety and Efficacy of C-CAR011 Treatment in Adult Subjects With r/r CD19+B-ALL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai AbelZeta Ltd. (Industry)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBMG2016003
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Relapsed or Refractory Acute Lymphoblastic Leukemia
Keywords: Relapsed or refractory acute lymphoblastic leukemia; Anti-CD19 chimeric antigen receptor T-cell
MeSH Terms: conditions — Recurrence; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- C-CAR011 (Experimental): In day 0, 1 and 2, CAR011 cells will be intravenous infused at the 10%, 30% and 60% ratio respectively.
  Interventions: Biological: C-CAR-011

INTERVENTIONS:
Biological: C-CAR-011 — CD19-targeted chimeric antigen receptor T cells
  Other Names: CAR-CD19

SUMMARY:
The trial is a single arm, single-center, non-randomized phase I clinical trial which is designed to evaluate the safety and efficacy of C-CAR011 in treatment of adult subjects with relapsed/refractory CD19+ B cells acute lymphoblastic leukemia(r/r CD19+B-ALL)

DETAILED DESCRIPTION:
This is a single-center, Open Label phase I clinical trial, 20 subjects planned to be enrolled. The trial have two stages (Phase I dose-escalation clinical trial and phase I dose expansion trial).Subjects will be divided into low-dose group, medium-dose group and high-dose group.Additional patients will be enrolled to confirm the optimal dose

Dose CAR+ cells/kg Low 0.5×106 Medium 1.5×106 High 3.0×106

ELIGIBILITY:
Inclusion Criteria:

* Age 14-75 years old, male or female.
* Volunteered to participate in this study and signed written informed consent form.
* Histologically diagnosed as CD19+B-ALL according to the NCCN Acute Lymphoblastic Leukemia Clinical Practice Guidelines (2016 version 1).
* Relapsed or refractory CD19+B-ALL (meet one of the following conditions)

  1. Refractory as defined not achieving a CR(complete remission, morphology<5% blasts) after two cycles of standard chemotherapy regimen.
  2. Duration of remission ≤ 12 months after the first induction chemotherapy regimen.
  3. Refractory disease after one or more salvage therapies.
  4. Two or more Bone Marrow relapse.
* Morphological disease in the bone marrow (≥ 5% blasts).
* Subjects with Philadelphia chromosome negative(Ph-) disease, or subjects with Philadelphia chromosome positive(Ph+) disease that are intolerant to or have failed 2 lines of tyrosine kinase inhibitor therapy (TKI), or if TKI therapy is contraindicated are eligible.
* No salvage chemotherapy therapy within 4 weeks prior to C-CAR011 therapy.
* No immunosuppressant(including but not limited to systemic corticosteroid therapy) within 4 weeks prior to C-CAR011 therapy.
* No antibody therapy within 4 weeks prior to C-CAR011 therapy.
* Normal cardiac function confirmed by ECHO with left ventricular ejection fraction (LVEF) ≧ 50%, no evidence of pericardial effusion and clinically significant arrhythmias.
* Baseline oxygen saturation ≧ 92% on room air and with normal pulmonary function, no evidence of active lung infection.
* No contraindications of peripheral blood apheresis.
* Expected survival ≧ 3 months.
* Eastern cooperative oncology group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* History of severe allergic disease or allergic to one or more drugs.
* Any kind of these laboratory testing: serum total bilirubin≧1.5mg/dl, serum albumin≦35g/L, ALT, AST≧2.5×ULN, serum creatinine≧2.0mg/dl, platelets≦50×109/L.
* Extramedullary disease.
* Relapsed disease after allogeneic hematopoietic stem cell transplantation.
* Diagnosis of Burkitt's leukemia/lymphoma according to WHO classification or chronic myelogenous leukemia lymphoid blast crisis.
* Subjects with concomitant genetic syndrome such as Fanconi anemia, Kostmann syndrome, Shwachman-Diamond syndrome or any other known bone marrow failure syndrome.
* Subjects with grade III or above severe hypertension(WHO/ISH Guidelines for the Management of Hypertension, 1999).
* History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months prior to enrollment.
* Subjects with class III and IV heart failure according to the NYHA Heart Failure Classifications;
* History of QT prolongation with clinically significant arrhythmias.
* History of epilepsy or other central nervous system disorders.
* History or presence of any central nervous system leukemia(CNS3, CNS4) disorder , with insensitive to intrathecal injection of or radiotherapy of head/spine; but effectively controlled cases will be eligible.
* Autoimmune diseases needing treatment, or immune deficiency or other diseases needing immunosuppressive therapy.
* Subjects with TKIs therapy (Ph+ ALL) within 1 week prior to enrollment.
* Severe active infection (uncomplicated urinary tract infections, bacterial pharyngitis allowed) or currently receiving intravenous antibiotic therapy and has received intravenous antibiotic therapy within one week. Prophylactic antibiotic, antiviral and antifungal treatment is permissible.
* Used any genetically modified T cell therapy.
* Presence of any indwelling line or drain (e.g., percutaneous nephrostomy tube, indwelling Foley catheter, biliary drain, or pleural/peritoneal/pericardial catheter). Ommaya reservoirs and dedicated central venous access catheters such as a Port-a-Cath or Hickman catheter are permitted.
* Live vaccine≦4 weeks prior to enrollment.
* Known infection with HIV, TB, hepatitis B (including carriers) or hepatitis C virus (anti-HCV positive).
* History of alcohol addiction , drug abuse or mental disease.
* Participated in any other clinical trial within three months prior to enrollment.
* Women who are pregnant or lactating or have breeding intent within 6 months.
* The investigators believe that any increase in the risk of the subject or interference with the results of the trial.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-08 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 30 days

SECONDARY OUTCOMES:
Overall response rate (ORR) | 8 weeks
Overall survival (OS) | 24 weeks
Minimal residual disease negative remission rate(MRD-) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Li Yu, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided